CLINICAL TRIAL: NCT01175343
Title: A Phase II Study of RO4929097 in Advanced Platinum Resistant Ovarian Cancer
Brief Title: RO4929097 in Treating Patients With Recurrent and/or Metastatic Epithelial Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03069; NCI-2012-03069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-079 (Other: University Health Network-Princess Margaret Hospital); 8635 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00071 (NIH); N01CM62201 (NIH); N01CM62203 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RO4929097) (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Blood and tumor tissue samples are collected for correlative studies. Ascitic fluid may also be collected.
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well RO4929097 works in treating patients with recurrent and/or metastatic epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the antitumor activity of RO4929097 in recurrent and / or metastatic epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer by progression free survival rate at the end of 4 cycles.

SECONDARY OBJECTIVES:

I. To assess the antitumor activity of RO4929097 through secondary endpoints including: overall response rate and CA125 response rate (GCIC criteria).

II. To assess the safety of single agent RO4929097 in advanced platinum resistant ovarian, fallopian tube and primary peritoneal cancers.

III. To explore expression of Notch biomarkers in advanced platinum resistant ovarian, fallopian, and primary peritoneal cancers.

IV. To explore the impact of RO49097 on ascitic fluid circulating tumor cells.

OUTLINE: This is a multicenter study.

Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and tumor tissue samples are collected for correlative studies. Ascitic fluid may also be collected.

After completion of study therapy, patients are followed up every month for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed ovarian epithelial carcinoma, fallopian tube carcinoma, or primary peritoneal carcinoma that is recurrent or metastatic; patients must have platinum resistant disease, as defined as treatment free interval less than 6 months post completion of platinum-based chemotherapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan

  * OR patients must have evidence of progression based on an elevated CA-125 (defined as a value of > 2 x ULN documented on two separate determinations made > 2 weeks apart, with the most recent being completed within 7 days prior to start of study treatment) if the physical exam is normal and maximum lesion diameter on the CT scan is < 20 mm with conventional techniques or as < 10 mm with spiral CT scan
* Patients must have completed any prior chemotherapy, radiotherapy or surgery >= 4 weeks (6 weeks for nitrosoureas or mitomycin C) before study entry

  * Prior radiotherapy is allowed provided that there is documented progression (either locally or systemically)
  * Patients may have had up to 2 prior lines of chemotherapy for recurrent or metastatic disease
  * Toxic effects from prior therapy must have resolved to grade 1 or less except for peripheral neuropathy and alopecia
* Life expectancy of greater than 12 weeks
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Patients must have normal organ and marrow function as defined below (within 7 days prior to start of study treatment):
* Hemoglobin >= 90 g/L
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 2.5 ULN (institutional upper limit of normal)
* AST (SGOT)/ALT (SGPT) =< 1.5 x institutional upper limit of normal (=< 5 times the ULN for patients with liver metastases)
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (using Cockcroft-Gault Formula)
* All radiology studies must be performed =< 4 weeks prior to the start of therapy
* No serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, psychiatric illness, or any other medical conditions that might be aggravated by treatment or limit compliance
* Currently no active, second malignancy other than non-melanoma skin cancers

  * NOTE: Patients are not considered to have a "current active" malignancy if they have completed anti-cancer therapy and are considered by their physician to be at less than 30% risk of relapse
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* The effects of RO4929097on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Notch signal pathway inhibitors are known to cause interruption of the embryonic signaling pathway and may lead to serious or life-threatening birth defects, including brain deformities, facial malformation, heart problems, or abnormal organs; if women of childbearing potential do not abstain* from sexual activity they must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry; women of childbearing potential can either be abstinent or use two forms of contraception for the duration of study participation and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she is participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately

  * Abstinent from sexual activity at least 4 weeks prior to study entry
  * Pregnancy Testing: Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator or clinical staff must confirm and document the patient's use of two contraceptive methods or abstinence, dates of negative pregnancy test, and confirm the patient's understanding of the potential of RO4929097 to cause serious or life-threatening birth defects
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
    * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin ®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; patients who are taking concurrent medications that are strong inducers, inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome, bowel obstruction, or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients who are serologically positive for Hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway inhibiting agent with the potential for serious or life-threatening birth defects or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Cardiovascular (within 7 days prior to start of study treatment): baseline QTc > 470 msec (female), QTc > 450 msec (male)

  * History of risk factors for QT interval prolongation, including, but not limited to family or personal history of long QT syndrome, recurrent syncope without known etiology or sudden unexpected death
  * History of torsade de pointes or other significant cardiac arrhythmias or the need for concomitant meds with known potential to prolong QT interval or antiarrhythmics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (12):
- United States (6):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
- Canada (6):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was taken off study prior to start of study drug for meeting exclusion criteria 3.2.5 (i.e. patient is taking concurrent medications that are strong inducers, inhibitors or substrates of CYP3A4 who cannot be switched to alternative medications).
Groups:
- Treatment (RO4929097): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Blood and tumor tissue samples are collected for correlative studies. Ascitic fluid may also be collected.
  Gamma-Secretase Inhibitor RO4929097: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (RO4929097)
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Four Cycle Progression-free Survival Rate
Description: Defined as the proportion of the study population that has not had tumor progression (symptomatic, RECIST progression, CA-125 progression) or died at the completion of the cycle four mark.
  RECIST criteria for progressive disease (PD) in target lesions: >= 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions is also considered progression. In non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
  CA-125 PD is based on the progressive serial elevation of serum CA-125 according to:
  A) elevated CA-125 pretreatment & normalization of CA-125 or C) CA-125 in normal range pretreatment: CA-125 >= 2x ULN on 2 occasions.
  B) elevated CA-125 pretreatment that never normalizes: CA-125 >= 2x nadir value on 2 occasions
Time Frame: 84 days (4 courses)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 44
Participants | 8

2. Secondary Outcome: Overall Response Rate
Description: Response was assessed by Response Evaluation Criteria In Solid Tumors (RECIST 1.1).
  Evaluation of Target Lesions:
  Complete response (CR) - disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response (PR) - at least 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Evaluation of Non-Target Lesions:
  Complete response (CR) - disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: Time from start of treatment to time of disease progression or death from any cause, whichever came first, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 44
Participants | 0

3. Secondary Outcome: CA125 Response Rate (GCIG Criteria)
Description: The CA-125 response rate is defined as the proportion of patients with a Gynecological Cancer Intergroup (GCIG) CA-125 response.
  CA-125 response is defined as the moment CA-125 is reduced by 50% from the last pre-treatment level prior to start of therapy. The response must be confirmed and maintained with a consecutive CA-125 for at least 28 days.
Time Frame: as for outcome 2
Population: There are 40 patients evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 40
Participants | 1

4. Secondary Outcome: Overall Survival
Description: Summary statistics, such as mean, median, counts and proportion, used to summarize the patients. Survival estimates computed using Kaplan-Meier method. Potential association between variables measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon rank sum tests may be substituted if necessary. Ninety-five percent confidence intervals will be constructed and selected results illustrated using figures and plots.
Time Frame: Up to 2 years
Population: 40 patients are evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 40
months | NA [NA to NA] — Not reached

5. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
Time Frame: Up to 2 years
Population: Adverse events analyzed include all serious adverse events (SAEs), and other (non-serious) treatment-related adverse events.There are 21 SAEs and 72 other (non-serious) adverse events.
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 44
Number analyzed (Adverse Events) | 93
Adverse Events
  All Adverse Events: Grade 1/2 | 71
  All Adverse Events: Grade 3/4 | 22
  Serious Adverse Events: number analyzed (Adverse Events) | 21
  Serious Adverse Events: Grade 1/2 | 2
  Serious Adverse Events: Grade 3/4 | 19
  Other Adverse Events: number analyzed (Adverse Events) | 72
  Other Adverse Events: Grade 1/2 | 69
  Other Adverse Events: Grade 3/4 | 3

6. Secondary Outcome: Expression of Notch Biomarkers in Advanced Platinum Resistant Ovarian, Fallopian, and Primary Peritoneal Cancers.
Description: An exploratory analysis for potential predictive biomarkers was performed on archival, paraffin-embedded tumor tissue for components of the Notch Pathway: Jagged-1 and NICD. The percentage of positive cells were scored into four categories: 0 (0%), 1 (1-33%), 2 (34-66%), and 3 (67-100%). The product of the intensity and percentage scores was used as the final score and classified as negative (0-4) or positive (5-9).
Time Frame: Up to 2 years
Population: 25 patients were assessed for Jagged-1 expression. 17 patients that were evaluable for response were assessed for NICD expression.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 25
Participants
  Jagged-1 expression: Positive | 23
  Jagged-1 expression: Negative | 2
  NICD expression: number analyzed (Participants) | 17
  NICD expression: Positive | 6
  NICD expression: Negative | 11

7. Secondary Outcome: Impact of RO49097 on Ascitic Fluid Circulating Tumor Cells
Description: Impact of RO49097 on ascitic fluid circulating tumor cells.
Time Frame: Up to 2 years
Population: Data were not collected.
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (RO4929097)
Serious Adverse Events (participants affected / at risk) | 10/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RO4929097) (N=44)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Parietal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (RO4929097) (N=44)
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 6
Anemia (Blood and lymphatic system disorders) | 5
Headache (Nervous system disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
ALT increase (Investigations) | 5
AST increase (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 3
Transient QT interval prolongation (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less